CLINICAL TRIAL: NCT05070351
Title: A Randomized Open-label Trial of Deprescribing Proton Pump Inhibitors to Reduce the Risk of Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt Creation
Brief Title: Deprescribing Proton Pump Inhibitors to Reduce Post-TIPS Hepatic Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00108517
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-03

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PPI deprescribing arm (Experimental): Patients taking a PPI (at least 20 mg omeprazole equivalent daily) will be instructed to stop taking their PPI.
  Interventions: Drug: PPI deprescribing
- PPI continuation arm (No Intervention): Patients will be instructed to continue taking their PPI (at least 20 mg omeprazole equivalent daily) as usual.

INTERVENTIONS:
Drug: PPI deprescribing — Patients currently on a proton pump inhibitor (PPI) undergoing transjugular intrahepatic portosystemic shunt (TIPS) creation as part of routine clinical care will be randomized to receive instructions to stop taking their PPI.
  Arms: PPI deprescribing arm

SUMMARY:
A total of 40 patients taking proton pump inhibitors (PPIs) who undergo transjugular intrahepatic portosystemic shunt (TIPS) creation as part of routine clinical care will be randomized in 1:1 fashion to either continue or discontinue their PPIs to determine whether these commonly used gastric acid suppressing agents increase risk of post-TIPS hepatic encephalopathy (HE). Patients will be assessed for symptoms of minimal HE (MHE), using the established psychometric hepatic encephalopathy score (PHES) battery of tests. MHE assessment will be conducted at two timepoints: at baseline prior to randomization and TIPS creation and approximately 4 weeks after randomization and TIPS creation. Stool samples will also be collected at both timepoints to allow characterization of the gastrointestinal (GI) tract microbiome using 16S rRNA sequencing. The pre to post-TIPS change in PHES scores will be compared between patients randomized to continue versus discontinue their PPIs. Quality of life (QOL) will also be assessed. Changes in the GI tract microbiome will be analyzed to determine whether this represents a potential biological mechanism linking PPI use with post-TIPS HE.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing TIPS creation as part of routine clinical care
* On PPIs therapy (at least 20 mg omeprazole equivalent daily)
* Provision of signed and dated informed consent form by participant or legal representative
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, age greater or equal to 18

Exclusion Criteria:

* Grade IV esophagitis or gastric or duodenal ulcer
* Recent endoscopic esophageal variceal band ligation necessitating PPI therapy for prevention of banding ulcer
* Zollinger-Ellison syndrome
* Active Helicobacter pylori infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Minimal hepatic encephalopathy | Approximately 6-8 weeks
  Minimal hepatic encephalopathy, as assessed by psychometric hepatic encephalopathy score

SECONDARY OUTCOMES:
Per-protocol evaluation of minimal hepatic encephalopathy | Approximately 6-8 weeks
  Minimal hepatic encephalopathy, as assessed by psychometric hepatic encephalopathy score, based on actual reported PPI use
Chronic liver disease specific quality of life | Approximately 6-8 weeks
  Chronic liver disease (CLDQ) specific QOL assessment
Gastroesophageal reflux specific quality of life | Approximately 6-8 weeks
  Gastroesophageal reflux (QOLRAD) specific QOL assessment
Overt hepatic encephalopathy | Approximately 6-8 weeks
  Episodes of overt hepatic encephalopathy (defined as West-Haven grade 2 or greater)
On-demand requirement for acid suppression therapy | Approximately 6-8 weeks
  Proportion of patients in the PPI discontinuation arm needing on-demand H2 blockers or PPIs for gastroesophageal reflux symptoms
Adverse events | Approximately 6-8 weeks
  Adverse events in the PPI continuation versus discontinuation arms

OTHER OUTCOMES:
Change in gastrointestinal tract microbiome | Approximately 6-8 weeks
  Pre-TIPS to post-TIPS change in stool taxon abundances as measured by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: James Ronald, MD PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT05070351/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT05070351/ICF_001.pdf